CLINICAL TRIAL: NCT00160420
Title: A Phase 2, 12-Month, Open Label Extension Study to Evaluate the Safety of J867(5 mg QD) in Subjects With Endometriosis
Brief Title: A Long-Term Study to Evaluate the Safety of Asoprisnil in the Treatment of Women With Endometriosis From Study M01-398
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Cynthia Mattia-Goldberg, Abbott
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M02-408
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2008-05-29 (Estimated); Status verified 2008-05

CONDITIONS: Endometriosis
Keywords: Pelvic pain; Dysmenorrhea; Dyspareunia; Infertility; asoprisnil
MeSH Terms: conditions — Endometriosis; Pelvic Pain; Dysmenorrhea; Dyspareunia; Infertility | interventions — asoprisnil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Asoprisnil

INTERVENTIONS:
Drug: Asoprisnil — 5mg Tablet, oral Daily for 12 months

SUMMARY:
The objective of this study is to determine the long-term safety of asoprisnil 5 mg for 12 months in women with endometriosis from study M01-398.

DETAILED DESCRIPTION:
Endometriosis, the presence of endometrial tissue outside the uterus, is a progressive, estrogen-dependent disease that occurs in menstruating women of reproductive age. Although all major endometriosis therapies are effective for the treatment of pain, no single treatment is superior to others in terms of efficacy. The major drawbacks of the current medical therapies are severe side effects such as hot flushes and osteoporosis. The objective of this study is to determine the long-term safety of asoprisnil 5 mg daily for 12 months in women with endometriosis, after an initial 12 weeks in study M01-398. The safety will be based on assessments of the endometrium, lipid profiles, adverse events, and changes from baseline laboratory values and vital signs.

ELIGIBILITY:
Inclusion Criteria:

* Completed 3 months of dosing and Month 3 procedures in study M01-398
* Otherwise in good health
* Month 3 (M01-398) ultrasound reveals no significant gynecologic disorder

Exclusion Criteria:

* Any abnormal lab or procedure result the study-doctor considers important
* Anticipated need for excluded hormonal therapy or unapproved narcotics

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2002-12; Primary Completion 2004-07 (Actual); Study Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in pelvic pain and dysmenorrhea assessed by visual analog scale. | Months 1,3,6,9,12 and final visit
Change from baseline in pelvic pain, dysmenorrhea, dyspareunia, pelvic tenderness and induration assessed by modified Biberoglu and Behrman grading scale. | Months 3,6,9,12 and final visit

SECONDARY OUTCOMES:
Percentage of subjects with amenorrhea. | Throught treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Chair — Abbott